CLINICAL TRIAL: NCT05313646
Title: Safety, Immunogenicity, and Batch Consistency of a Single Dose of a Recombinant Adenovirus Type-5-vectored COVID-19 Vaccine in Chinese Healthy Adults Aged 18 Years and Above: a Randomized, Double-blind, Parallel-controlled Clinical Trial
Brief Title: Clinical Evaluation for Batch Consistency of Ad5-nCoV in Chinese Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT111
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 Vaccine; Batches consistency; Adenovirus type-5-vectored; Safety; Immunogenicity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Subjects in adults cohort and elderly cohort will be randomized in a 1:1:1 ratio to receive one of three consecutive batches of Convidecia, respectively.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and investigators will be kept blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- batch 1 of Ad5-nCoV (Experimental): Eligible subjects in both cohort were vaccinated with one injection of Ad5-nCoV, lot NCOV202101001.
  Interventions: Biological: batch 1 of Ad5-nCoV
- batch 2 of Ad5-nCoV (Experimental): Eligible subjects in both cohort were vaccinated with one injection of Ad5-nCoV, lot NCOV202101002.
  Interventions: Biological: batch 2 of Ad5-nCoV
- batch 3 of Ad5-nCoV (Experimental): Eligible subjects in both cohort were vaccinated with one injection of Ad5-nCoV, lot NCOV202102003.
  Interventions: Biological: batch 3 of Ad5-nCoV

INTERVENTIONS:
Biological: batch 1 of Ad5-nCoV — The vaccine is a replication defective Ad5 vectored vaccine expressing the full-length spike glycoprotein of SARS-CoV-2 produced by CanSino, lot NCOV202101001. It contains 5×10^10 viral particles per 0.5 mL in a vial.
  Other Names: Convidecia
  Arms: batch 1 of Ad5-nCoV
Biological: batch 2 of Ad5-nCoV — The vaccine is a replication defective Ad5 vectored vaccine expressing the full-length spike glycoprotein of SARS-CoV-2 produced by CanSino, lot NCOV202101002. It contains 5×10^10 viral particles per 0.5 mL in a vial.
  Other Names: Convidecia
  Arms: batch 2 of Ad5-nCoV
Biological: batch 3 of Ad5-nCoV — The vaccine is a replication defective Ad5 vectored vaccine expressing the full-length spike glycoprotein of SARS-CoV-2 produced by CanSino, lot NCOV202102003. It contains 5×10^10 viral particles per 0.5 mL in a vial.
  Other Names: Convidecia
  Arms: batch 3 of Ad5-nCoV

SUMMARY:
This is a randomized, double-blind, parallel-controlled, equivalence trial, for evaluation of safety and immunogenicity, and batch-to-batch consistency of a recombinant adenovirus type-5-vectored Covid-19 vaccine Convidecia in one shot schedule in Chinese healthy adults aged 18 years and above. In total 1050 healthy adults will be recruited in this study. Subjects in both cohort will be randomized stratified into two cohort by age(18~59 years and≥60 years) in a 1:1:1 ratio to receive one of three consecutive batches of Convidecia. The primary objective is to test the equivalence of the immune responses to three consecutive manufacturing lots of Convidecia in healthy adults. The secondary objectives were to evaluate the immunogenicity and safety of Convidecia for each lot and the pooled data of three lots)

ELIGIBILITY:
Inclusion Criteria:

1. healthy participants aged 18 years and above who have not received COVID-19 vaccine.
2. The subjects can provide with informed consent and sign informed consent form (ICF).

4. The subjects are able to and willing to comply with the requirements of the clinical trial program and could complete the follow-up of the study.

5. Axillary temperature ≤ 37.0℃. 6. negative IgM and IgG against SARS-CoV-2 7. with BMI between18.5 to 30.0 8. No history of epidemiological contact with COVID-2019 9. have not been to medium or high risk areas in the past 21 days and have no history of departure.

10. be determined to be healthy by medical history, physical examination and clinical examination and meet the requirements for immunization of this product.

Exclusion criteria:

1. Medical history or family history of convulsion, epilepsy, encephalopathy and psychosis.
2. Allergic to any component of the research vaccines, or a history of hypersensitivity or serious reactions to vaccination.
3. Women with positive urine pregnancy test, pregnant or breast-feeding, or have a pregnancy plan in this study.
4. Suffering from acute febrile disease, infectious disease, or SARS infection history
5. Serious cardiovascular disease, such as arrhythmia, conduction block, myocardial infarction, severe hypertension, which cannot be controlled by medication (systolic blood pressure ≥180mmHg, diastolic blood pressure ≥110mmHg)
6. Have severe chronic diseases or unstable condition ( Grade 3 or higher as defined in the guidelines for the classification of adverse events in clinical trials for prophylactic vaccines), Such as diabetes, thyroid disease and so on.
7. Congenital or acquired angioedema / neuroedema.
8. had urticaria one year before this vaccination.
9. Asplenia or functional asplenia.
10. Thrombocytopenia or other clotting disorder (this may contraindicate intramuscular injection).
11. Faintng during acupuncture treatment
12. Received immunosuppressant therapy, antiallergic therapy, cytotoxic therapy, high dose inhaled corticosteroid over the past 6 months (excluding corticosteroid spray for allergic rhinitis, surface corticosteroid for acute non-complicated dermatitis, and corticosteroid with dose less than 20mg/ day)
13. Received blood products within 4 months before vaccination.
14. Received other investigational drugs within 1 month prior to receiving the investigational vaccines.
15. Received other live attenuated vaccines within 1 month prior to receiving the investigational vaccines.
16. Received subunit or inactivated vaccine within 14 days prior to receiving investigational vaccine.
17. Be receiving anti-tuberculosis treatment
18. Have the history of SARS-CoV-2 infection or COVID-19
19. Any medical, psychological, social or other conditions that, in the investigator's judgment, are inconsistent with the study protocol or affect the subjects' informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
GMTs of SARS-CoV-2 RBD-specific binding IgG on day 28 after vaccination. | On day 28 after vaccination
  GMTs of SARS-CoV-2 RBD-specific binding IgG on day 28 after vaccination.

SECONDARY OUTCOMES:
GMFIs of SARS-CoV-2 RBD-specific binding IgG on day 28 after vaccination. | On day 28 after vaccination
  GMFIs of SARS-CoV-2 RBD-specific binding IgG on day 28 after vaccination.
Propotion of participants with at least four-fold increase of post-vaccination antibody level against SARS-CoV-2 RBD-specific binding IgG compared to that at baseline on day 28 after vaccination. | On day 28 after vaccination
  Propotion of participants with at least four-fold increase of post-vaccination antibody level against SARS-CoV-2 RBD-specific binding IgG compared to that at baseline on day 28 after vaccination.
GMTs of SARS-CoV-2 RBD-specific binding IgG on day 28 after vaccination stratified by neutralizing antibody levels against Ad5 at baseline. | On day 28 after vaccination
  GMTs of SARS-CoV-2 RBD-specific binding IgG on day 28 after vaccination stratified by neutralizing antibody
Incidence of solicited adverse events within 7 days after vaccination. | Within 7 days after vaccination
  Incidence of solicited adverse events within 7 days after vaccination.
Incidence of adverse reactions within 28 days after vaccination. | Within 28 days after vaccination
  Incidence of adverse reactions within 28 days after vaccination.
Incidence of unsolicited adverse events within 28 days after vaccination. | Within 28 days after vaccination
  Incidence of unsolicited adverse events within 28 days after vaccination.
Incidence of serious adverse events (SAE) within the 6 months after vaccination. | Within the 6 months after vaccination
  Incidence of serious adverse events (SAE) within the 6 months after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, MSc, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Guanyun Center for Disease Control and Prevention, Lianyungang, Jiangsu, China

REFERENCES:
- [Derived] Li ZP, Shi YF, Hou LH, Jin PF, Ma SH, Pan HX, Zhang JL, Shan YM, Huang HT, Wu SP, Du P, Wang X, Wang LL, Wang RJ, Wang Y, Wang XW, Zhu FC, Li JX. Batch-to-batch consistency trial of an adenovirus type-5 vector-based COVID-19 vaccine in adults aged 18 years and above. Expert Rev Vaccines. 2022 Dec;21(12):1843-1849. doi: 10.1080/14760584.2022.2119133. Epub 2022 Sep 1. PMID 36048417